CLINICAL TRIAL: NCT03873480
Title: Administration of Local Anesthetic in Trigger Thumb Surgery: A Randomized Clinical Trial
Brief Title: Trigger Thumb Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-015288
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Trigger Thumb
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): Participants randomized into the intervention group will receive an injection of 2.5 cc of 0.25% marcaine without epinephrine prior to the incision. The local anesthetic will be administered by the treating surgeon. All other aspects of the procedure will be kept in accordance with the standard of care for trigger thumb surgeries.
  Interventions: Procedure: Administration of Marcaine without Epinephrine prior to the start of surgery
- Non-Intervention Arm (No Intervention): Those that are not randomized into the intervention group will receive the standard of care for a trigger thumb release, which is administration of 2.5 cc of 0.25% marcaine without epinephrine following completion of surgery. The local anesthetic will be administered by the treating surgeon.

INTERVENTIONS:
Procedure: Administration of Marcaine without Epinephrine prior to the start of surgery — The intervention is the timing of administration of marcaine without epinephrine during a trigger thumb surgery.
  Arms: Intervention Arm

SUMMARY:
We are conducting this study to determine if administration of local anesthetic to the thumb prior to surgery can reduce the amount of anesthetic gas given during the course of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 0-4 years, presenting to the Children's Hospital of Philadelphia (CHOP) Department of Orthopaedics with unilateral trigger thumb that requires surgical treatment.
2. American Society of Anaesthesiologists (ASA) Classification of 1 or 2.
3. Parental/guardian permission (informed consent).

Exclusion Criteria:

1. Males or females over the age of 4.
2. ASA Classification higher than 2.
3. Patients presenting with systemic diseases or significant comorbidities.
4. Patients that received treatment for trigger thumb at an outside institution.

Ages: 0 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Difference in administered anesthesia | 3 years
  The primary outcome will be the difference in administered gaseous sevoflurane during the course of trigger thumb surgery between the control group and intervention group.

SECONDARY OUTCOMES:
Difference in observed pain score | 3 years
  The secondary outcome will be the difference in observed pain scores during the post-operative period following a trigger thumb surgery between the control group and intervention group. The FLACC (face, legs, activity, consolability) Behavioural pain scale will be used. There are 5 components, e.g. face, legs, activity, cry, and consolability, that are given a grade of 0, 1, or 2. The sum of the each component grade will give the pain scale score.
  0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 = Moderate pain 7-10 = Severe discomfort/pain
Difference in operative time | 3 years
  The secondary outcome will be the difference in operative time during the course of a trigger thumb surgery between the control group and intervention group.
Difference in length of stay | 3 years
  The secondary outcome will be the difference in total length of study following a trigger thumb surgery between the control group and intervention group.
Difference in complication rates | 3 years
  The secondary outcome will be the difference in complication rates following a trigger thumb surgery between the control group and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Apurva S Shah, MD, MBA, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual participant data will not be made available.